CLINICAL TRIAL: NCT05590377
Title: A Phase 1/2a Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Modakafusp Alfa in Combination With Daratumumab Subcutaneous in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Modakafusp Alfa Together With Daratumumab Adults With Relapsed or Refractory Multiple Myeloma
Acronym: iinnovate-3
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: After completion of Phase 1 Dose Escalation of this study the sponsor decided not to proceed with Phase 2a due to strategic reasons. Thus, no participants were enrolled for Phase 2a and the study was terminated early.
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-573-2001; 2022-002169-14 (EudraCT Number)
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab (Experimental): Modakafusp alfa 80 mg, infusion, intravenously (IV), once every 4 weeks (Q4W) with daratumumab 1800 mg, subcutaneously (SC), once weekly (QW) in Cycles 1 and 2, twice weekly (Q2W) in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression.
  Interventions: Drug: Modakafusp Alfa; Drug: Daratumumab
- Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab (Experimental): Modakafusp alfa 120 mg, infusion, IV, Q4W with daratumumab 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression.
  Interventions: Drug: Modakafusp Alfa; Drug: Daratumumab
- Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab (Experimental): Modakafusp alfa 240 mg, infusion, IV, Q4W with daratumumab 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression.
  Interventions: Drug: Modakafusp Alfa; Drug: Daratumumab
- Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab (Experimental): Modakafusp alfa at dose level 1 (DL1) [selected from Phase 1 Dose Escalation] with daratumumab SC 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression.
  Interventions: Drug: Modakafusp Alfa; Drug: Daratumumab
- Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab (Experimental): Modakafusp alfa at dose level 2 (DL2) [selected from Phase 1 Dose Escalation] with daratumumab SC 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression.
  Interventions: Drug: Modakafusp Alfa; Drug: Daratumumab

INTERVENTIONS:
Drug: Modakafusp Alfa — Modakafusp alfa intravenous infusion
  Other Names: TAK-573
Drug: Daratumumab — Daratumumab SC injection

SUMMARY:
The main aim of this study is to determine safety and tolerability of modakafusp alfa given together with daratumumab to find out the best treatment dose. Another aim of this study is to learn more about the characteristics of modakafusp alfa.

DETAILED DESCRIPTION:
The drug being tested in this study is called modakafusp alfa (TAK-573). Modakafusp alfa is being tested to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary efficacy in combination with daratumumab in participants with relapsed or refractory multiple myeloma (RRMM). The study will consist of 2 phases: Phase 1 Dose Escalation and a Phase 2a Dose Finding.

The study will enroll approximately 58 patients. Approximately 18 participants will be enrolled in the Phase 1 Dose Escalation/De-escalation and two dose levels of modakafusp alfa in combination with daratumumab SC will be selected to be further explored in the randomized Phase 2a Dose Finding part of the study wherein, approximately 40 participants will be randomly assigned by chance (like flipping a coin) to one of the two treatment groups:

* Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab
* Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 60 months. Participants who discontinue study drug treatment for reasons other than progressive disease will continue progression-free survival (PFS) follow-up every 4 weeks from the end of treatment (EOT) visit until the occurrence of progressive disease, death, the start of subsequent systemic antineoplastic therapy, study termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Documented multiple myeloma (MM) diagnosis per IMWG criteria.
2. Measurable disease, defined as at least 1 of the following:

   1. Serum M protein ≥0.5 grams per deciliter [g/dL] (≥5 g/L) on serum protein electrophoresis (SPEP).
   2. Urine M protein ≥200 mg/24 hours on urine protein electrophoresis (UPEP).
   3. Serum free light chain (FLC) assay with involved FLC level ≥10 mg/dL (≥100 mg/L) provided serum FLC ratio is abnormal.
3. For participants in the Phase 1 Dose Escalation only:

   Must have received at least 3 prior lines of therapy, including at least 1 proteosome inhibitor (PI), 1 immunomodulatory imide drug (IMiD), and 1 anti-CD38 monoclonal antibody (mAb) drug; or who are triple refractory to a PI, an IMiD, and an anti-CD38 mAb drug, regardless of the number of prior line(s) or therapy.
4. For participants in Phase 2a Dose Finding only:

   1. Received 1 to 3 prior line(s) of antimyeloma therapy.
   2. Must be refractory to prior lenalidomide treatment.
   3. Participants must be sensitive (nonrefractory) or naïve to prior anti-CD38 mAb treatment.
   4. Documented progressive disease on or after the last regimen.
   5. Participants must have PR or better to at least 1 line of prior therapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at screening.

Exclusion Criteria:

1. Prior exposure to modakafusp alfa.
2. Participant has polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, solitary plasmacytoma, amyloidosis, Waldenström macroglobulinemia, plasma cell leukemia, or lymphoplasmacytic lymphoma.
3. Participant has not recovered from adverse reactions to prior myeloma treatment or procedures (chemotherapy, immunotherapy, radiation therapy) to NCI CTCAE, Version 5 Grade ≤1 or baseline, except for alopecia.
4. Previous allogeneic stem cell transplant at any time or autologous stem cell transplant (ASCT) within 12 weeks of planned start of dosing.
5. Seropositive for hepatitis B, or known history of seropositivity for hepatitis C or of seropositivity for human immunodeficiency virus (HIV).
6. Participant has congestive heart failure (New York Heart Association Grade ≥II), cardiac myopathy, active ischemia, or any other uncontrolled cardiac condition such as angina pectoris, clinically significant arrhythmia requiring therapy including anticoagulants, or clinically significant uncontrolled hypertension.
7. Participant has QT interval corrected by the Fridericia method >480 milliseconds [msec] (Grade ≥2).
8. Participant has a chronic condition that will require the chronic use of systemic corticosteroids >10 milligrams per day (mg/d) of prednisone or equivalent on top of any required corticosteroids for multiple myeloma (MM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (13):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Fort Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - HCA Midwest Health (Midwest Ventures Group HCA MidAmerica Division), Overland Park, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Summit Medical Group PA, Florham Park, New Jersey
  - New York Cancer and Blood Specialists, Bay Shore, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - University of Cincinnati - Vontz Center for Molecular Studies, Cincinnati, Ohio
  - Tranquil Clinical Research, Webster, Texas
- Australia (2):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Centre Hospitalier Universitaire De Sherbrooke (CHUS) - Centre de Recherche Clinique Etienne-Le Bel (CRCELB) Hopital Fleurimont, Sherbrooke, Quebec, Canada
- China (4):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Wuhan Union Hospital, Wuhan, Hubei
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality
  - Zhejiang University School of Medicine - The First Affiliated Hospital (Zhejiang Provincial First Hospital), Hangzhou, Zhejiang
- France (2):
  - CHRU Lille, Lille, Hauts-de-France
  - Institut Paoli-Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
- South Korea (3):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Fundacion Instituto de Estudios Ciencias de la Salud de Castilla y Leon-Investigacion Biomedica de Salamanca (IBSAL), Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites globally from 23 January 2023 to 22 May 2024.
Pre-assignment Details: Participants with multiple myeloma were enrolled in Phase 1 (Dose Escalation) to receive modakafusp alfa (80 milligrams [mg], 120 mg or 240 mg) + daratumumab. No participants were enrolled in Phase 2a (Dose Finding) as the study was terminated by the Sponsor due to strategic reasons.
Groups:
- Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab: Participants received modakafusp alfa 80 mg, infusion, IV, Q4W with daratumumab 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression or up to 60 weeks.
- Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab: Participants received modakafusp alfa 120 mg, infusion, IV, Q4W with daratumumab 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression or up to 48 weeks.
- Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab: Participants received modakafusp alfa 240 mg, infusion, IV, Q4W with daratumumab 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression or up to 36 weeks.
- Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab: Participants were planned to receive modakafusp alfa at dose level 1 (DL1) [selected from Phase 1 Dose Escalation] with daratumumab SC 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression.
- Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab: Participants were planned to receive modakafusp alfa at dose level 2 (DL2) [selected from Phase 1 Dose Escalation] with daratumumab SC 1800 mg, SC, QW in Cycles 1 and 2, Q2W in Cycles 3 to 6, and Q4W thereafter in each 28-day treatment cycle until disease progression.
Period: Overall Study
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Started | 3 | 6 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 6 | 0 | 0
Not completed — Death | 1 | 1 | 2 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 5 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received at least 1 dose, even an incomplete dose, of any study drug. After completion of Phase 1 Dose Escalation of this study the sponsor decided not to proceed with Phase 2a due to strategic reasons. Thus, no participants enrolled in Phase 2a and it is therefore not presented here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab | Total
Number analyzed (Participants) | 3 | 6 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (18.34) | 63.7 (11.64) | 59.2 (12.02) | 63.5 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 1 | 4 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 4 | 3 | 10
  Unknown or Not Reported | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 3 | 0 | 1 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLT)
Description: DLT was defined as any of the treatment-emergent adverse events (TEAEs) that occurred during Cycle 1 and were considered by the investigator to be at least possibly related to modakafusp alfa. Toxicity was evaluated according to national cancer institute common terminology criteria for adverse events (NCI CTCAE) Version 5.0.
Time Frame: Phase 1: Cycle 1 (cycle length=28 days)
Population: The Dose Limiting Toxicity (DLT)-evaluable Population included all participants from the Phase 1 dose escalation portion who experienced a DLT in Cycle 1 in the treatment phase of the study or had completed the Cycle 1 dose of modakafusp alfa and at least 75% of the planned dose of daratumumab SC.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab
Number analyzed (Participants) | 3 | 6 | 6
Participants | 0 | 0 | 1

2. Primary Outcome: Phase 1: Number of Participants Reporting One or More TEAEs and Per Severity
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Severity grades for TEAEs were evaluated as per the NCI CTCAE Version 5.0.
Time Frame: Phase 1: Up to 15.9 months
Population: The Safety Population included all participants who received at least 1 dose, even an incomplete dose, of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab
Number analyzed (Participants) | 3 | 6 | 6
Participants
  Grade 1 | 1 | 0 | 0
  Grade 2 | 0 | 2 | 1
  Grade 3 | 2 | 4 | 3
  Grade 4 | 0 | 0 | 1
  Grade 5 | 0 | 0 | 1

3. Primary Outcome: Phase 2a: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve a confirmed partial response (PR) or better during the study in the safety population. ORR will be assessed by the investigator per International Myeloma Working Group (IMWG) criteria.
Time Frame: Phase 2a: Up to 15.9 months
Population: After completion of Phase 1 Dose Escalation of this study the sponsor decided not to proceed with Phase 2a due to strategic reasons. Thus, no participants were enrolled for Phase 2a and no data was collected for this outcome measure due to study termination.
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 1: Cmax: Single-Dose Maximum Observed Serum Concentration for Modakafusp Alfa
Time Frame: Phase 1: Days 1, 8, 15, and 22 of Cycles 1 and 2: Pre-dose, and at multiple time points up to 4 hours post-dose; Day 2 of Cycles 1 and 2: Post-dose (cycle length=28 days)
Reporting Status: Not Posted

5. Secondary Outcome: Phase 1: Tmax: Time to First Occurrence of Maximum Serum Concentration (Cmax) for Modakafusp Alfa
Time Frame: as for outcome 4
Reporting Status: Not Posted

6. Secondary Outcome: Phase 1: AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for Modakafusp Alfa
Time Frame: as for outcome 4
Reporting Status: Not Posted

7. Secondary Outcome: Phase 1: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration
Time Frame: as for outcome 4
Reporting Status: Not Posted

8. Secondary Outcome: Phase 1: Apparent Serum Terminal Disposition Rate Constant for Modakafusp Alfa
Time Frame: as for outcome 4
Reporting Status: Not Posted

9. Secondary Outcome: Phase 1: Apparent Serum Terminal Disposition Phase Half-life for Modakafusp Alfa
Time Frame: as for outcome 4
Reporting Status: Not Posted

10. Secondary Outcome: Phase 1: Total Clearance After Intravenous Administration for Modakafusp Alfa
Time Frame: as for outcome 4
Reporting Status: Not Posted

11. Secondary Outcome: Phase 1: Volume of Distribution at Steady State After Intravenous (IV) Administration for Modakafusp Alfa
Time Frame: as for outcome 4
Reporting Status: Not Posted

12. Secondary Outcome: Phase 1: Cmax: Single-Dose Maximum Observed Serum Concentration for Daratumumab
Time Frame: as for outcome 4
Reporting Status: Not Posted

13. Secondary Outcome: Phase 1: Tmax: Time to First Occurrence of Maximum Serum Concentration (Cmax) for Daratumumab
Time Frame: as for outcome 4
Reporting Status: Not Posted

14. Secondary Outcome: Phase 1: Ctrough: Single-Dose and Multiple-dose Observed Concentration at the End of a Dosing Interval for Daratumumab
Time Frame: as for outcome 4
Reporting Status: Not Posted

15. Secondary Outcome: Phase 1: AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for Daratumumab
Time Frame: as for outcome 4
Reporting Status: Not Posted

16. Secondary Outcome: Phase 1: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for Daratumumab
Time Frame: as for outcome 4
Reporting Status: Not Posted

17. Secondary Outcome: Phase 1: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a confirmed PR or better during the study in the safety population. ORR will be assessed by the investigator per IMWG criteria.
Time Frame: Phase 1: Up to 15.9 months
Population: The Response-evaluable Population included all participants who received at least 1 dose, even an incomplete dose, of any study drug, have a disease assessment at screening (baseline evaluation), and at least 1 postbaseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab
Number analyzed (Participants) | 3 | 6 | 6
percentage of participants | 33.3 [0.84 to 90.57] | 66.7 [22.28 to 95.67] | 50.0 [11.81 to 88.19]

18. Secondary Outcome: Phase 1 and Phase 2a: Duration of Response (DOR)
Description: DOR is defined as the time from the date of first documentation of a confirmed PR or better to the date of first documentation of confirmed progressive disease or death due to any cause, whichever occurs first. DOR will be calculated for confirmed responders only (PR or better). DOR will be assessed by the investigator as per IMWG criteria.
Time Frame: Up to 15.9 months
Reporting Status: Not Posted

19. Secondary Outcome: Phase 1 and Phase 2a: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose administration of any study drug to the first documentation of confirmed progressive disease or death due to any cause, whichever occurs first. PFS will be assessed by the investigator as per IMWG criteria.
Time Frame: Up to 15.9 months
Reporting Status: Not Posted

20. Secondary Outcome: Phase 1 and Phase 2a: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose administration of any study drug to the documentation of death due to any cause. OS will be assessed by the investigator as per IMWG criteria.
Time Frame: Up to 15.9 months
Reporting Status: Not Posted

21. Secondary Outcome: Phase 1 and Phase 2a: Number of Participants With Anti-drug Antibodies (ADA)
Description: After completion of Phase 1 Dose Escalation of this study the sponsor decided not to proceed with Phase 2a due to strategic reasons and hence no participants were enrolled for Phase 2a.
Time Frame: Up to 15.9 months
Population: Immunogenicity-evaluable Population included participants who received at least 1 dose of modakafusp alfa in combination with daratumumab SC (partial or complete) with a baseline assessment & at least 1 postbaseline immunogenicity assessment. No data was collected for this outcome measure due to study termination. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab
Number analyzed (Participants) | 3 | 6 | 0
Participants | 3 | 2 | 0

22. Secondary Outcome: Phase 1 and Phase 2a: Titer of Anti-drug Antibodies
Time Frame: Up to 15.9 months
Reporting Status: Not Posted

23. Secondary Outcome: Phase 1 and Phase 2a: Number of Participants With Neutralizing Antibodies (NAb) Against Study Drug
Time Frame: Up to 15.9 months
Reporting Status: Not Posted

24. Secondary Outcome: Phase 1 and Phase 2a: Rate of Measurable [Minimal] Residual Disease Negative (MRD[-]) Complete Response (CR)
Description: MRD[-] CR rate is defined as the percentage of participants who achieve confirmed CR assessed by the investigator and MRD[-] status using a threshold of 10^-5. The analysis will be based on the response-evaluable population. No participants had sCR or CR in Phase 1 thus the overall number of participants analyzed is zero.
Time Frame: Up to 15.9 months
Population: Only participants who had a confirmed stringent CR (sCR) or complete response (CR) were to be analyzed for this outcome measure. After completion of Phase 1 Dose Escalation of this study the sponsor decided not to proceed with Phase 2a due to strategic reasons. Thus, no participants were enrolled for Phase 2a & no data was collected for this outcome measure due to study termination.
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Phase 1 and Phase 2a: Duration of Measurable [Minimal] Residual Disease (MRD) Negativity
Description: Duration of MRD negativity for participants achieving MRD negativity is defined as the time from the date of first documentation of MRD negativity to the first documentation of MRD positivity or confirmed progressive disease, whichever occurs first. It will be calculated for participants achieving MRD negativity only. No participants had sCR or CR in Phase 1 thus the overall number of participants analyzed is zero.
Time Frame: Up to 15.9 months
Population: as for outcome 24
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Phase 2a: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants who had a confirmed response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), or minimal response based on investigators' disease assessment per IMWG criteria.
Time Frame: Phase 2a: Up to 15.9 months
Population: After completion of Phase 1 Dose Escalation of this study the sponsor decided not to proceed with Phase 2a due to strategic reasons. Thus, no participants were enrolled for Phase 2a & no data was collected for this outcome measure due to study termination.
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Phase 2a: Duration of Clinical Benefit (DCB)
Description: DCB is defined as the time from the date of first documentation of a minimal response or better to the date of first documentation of confirmed progressive disease or death due to any cause, whichever occurs first. DCB will be calculated for only participants who achieved a minimal response or better. DCB will be assessed by the investigator as per IMWG criteria.
Time Frame: Phase 2a: Up to 15.9 months
Population: After completion of Phase 1 Dose Escalation of this study the sponsor decided not to proceed with Phase 2a due to strategic reasons (no safety concerns). Thus, no participants were enrolled for Phase 2a & no data was collected for this outcome measure due to study termination.
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Phase 2a: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a confirmed response of sCR, CR, VGPR, PR, minimal response, or stable disease (SD) based on investigators' disease assessment per IMWG criteria.
Time Frame: Phase 2a: Up to 15.9 months
Population: as for outcome 27
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Phase 2a: Duration of Disease Control
Description: Duration of disease control is defined as the time from date of first documentation of SD or better to the date of first documentation of confirmed progressive disease or death due to any cause. Duration of disease control will be calculated for only patients who achieved SD or better. It will be assessed by the investigator per IMWG criteria.
Time Frame: Phase 2a: Up to 15.9 months
Population: as for outcome 27
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Phase 2a: Time to Progression (TTP)
Description: TTP is defined as the time from the date of randomization to the first documentation of confirmed progressive disease as defined by IMWG criteria, assessed by the investigator. Participants without documentation of confirmed progression will be censored at the date of last adequate disease assessment. The analysis will be based on the intent-to-treat (ITT) population.
Time Frame: Phase 2a: Up to 15.9 months
Population: as for outcome 27
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Phase 2a: Time to Response (TTR)
Description: TTR is defined as time from the date of first dose administration of any study drug to the date of the first documentation of a confirmed PR or better. TTR will be calculated for responders only. TTR will be assessed by the investigator per IMWG criteria.
Time Frame: Phase 2a: Up to 15.9 months
Population: as for outcome 27
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Phase 2a: Time to Next Treatment (TTNT)
Description: TTNT is defined as the time from the date of first dose administration of any study drug to the date of the first dose initiation of the next line of anticancer therapy for any reason or death from any cause, whichever comes first. Participants who have not started the next-line therapy will be censored at the date last known to be alive before subsequent anticancer therapy.
Time Frame: Phase 2a: Up to 15.9 months
Population: as for outcome 27
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Phase 2a: Number of Participants Reporting One or More TEAEs and Per Severity
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Severity grades for TEAEs will be evaluated as per the NCI CTCAE Version 5.0.
Time Frame: Phase 2a: Up to 15.9 months
Population: as for outcome 27
Arm/Group | Phase 2a Dose Finding: Modakafusp Alfa (DL1) + Daratumumab | Phase 2a Dose Finding: Modakafusp Alfa (DL2) + Daratumumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Phase 1: Up to 15.9 months
Description: The Safety Population was defined as all participants who received at least 1 dose, even an incomplete dose, of any study drug. The sponsor decided not to proceed with Phase 2a after phase 1 completion due to strategic reasons. Thus, no participants were enrolled & no adverse events were reported for Phase 2a.
Arm/Group | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/6 | 2/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab (N=3) | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab (N=6) | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab (N=6)
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Dose Escalation) Modakafusp Alfa 80 mg + Daratumumab (N=3) | Phase 1 (Dose Escalation) Modakafusp Alfa 120 mg + Daratumumab (N=6) | Phase 1 (Dose Escalation) Modakafusp Alfa 240 mg + Daratumumab (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Dry eye (Eye disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 2
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 2
Rash pustular (Infections and infestations) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT05590377/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT05590377/SAP_001.pdf